CLINICAL TRIAL: NCT07304167
Title: Investigation of the Effectiveness of a Video-Based Exercise (Exergame) Program in Women With Fibromyalgia: A Randomized Controlled Trial
Brief Title: Investigation of the Effectiveness of a Exergame Program in Women With Fibromyalgia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Halic University (Other)
Responsible Party: Principal Investigator, Ayşenur Çetinkaya, PT, PhD, Halic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Acetinkaya007
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Fibromyalgia; Exergaming
Keywords: Fibromyalgia; Exergaming; Exercise; Rehabilitation
MeSH Terms: conditions — Fibromyalgia; Motor Activity | interventions — Exergaming

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exergame group (Experimental): Participants in this group will perform exergame-based exercises.
  Interventions: Other: Exergaming
- Home-based exercise group (Experimental): Participants in this group will perform home-based exercise sessions.
  Interventions: Other: Home-based exercise

INTERVENTIONS:
Other: Exergaming — Participants in the exergame group will perform exercises using the Nintendo Switch game Ring Fit Adventure under the supervision of a physiotherapist, twice a week for four weeks. The exergame program was designed by a specialist physiotherapist.
  Arms: Exergame group
Other: Home-based exercise — Participants in the home-based exercise group will perform exercises prescribed by a specialist physiotherapist as a home program, twice a week for four weeks. The exercises will be taught to participants in face-to-face sessions. Once a week, participants in the home-based exercise group will meet via Zoom to monitor exercise accuracy and progression. The home-based exercise program was adapted from the study conducted by Gentile et al. (2024).
  Arms: Home-based exercise group

SUMMARY:
The goal of this clinical trial is to compare the effects of an exergame-based exercise program and a home-based exercise program in women aged 30-70 years diagnosed with fibromyalgia (FM).

The main questions it aims to answer are:

Does an exergame-based program using the Nintendo Switch game Ring Fit Adventure improve pain, balance, and functional mobility in women with fibromyalgia? Is the exergame program more effective than a traditional home-based exercise program in improving physical and psychosocial outcomes? Researchers will compare the exergame group and the home-based exercise group to determine whether game-based exercises provide superior benefits in pain reduction, balance, and quality of life.

Participants will:

Be randomly assigned to either the exergame or the home-based exercise group. Exercise twice a week for four weeks under the supervision of a physiotherapist or via remote monitoring.

Undergo evaluations before and after the 4-week training period, and again after a 4-week detraining period.

Assessments will include:

Pain intensity (Visual Analog Scale) Disease severity (Revised Fibromyalgia Impact Questionnaire, Widespread Pain Index, Symptom Severity Scale, Fibromyalgia Severity Scale) Lower extremity strength (Sit-to-Stand Test) Functional mobility (Timed Up and Go Test) Balance (Single-Leg Stance Test, Berg Balance Scale) Psychosocial status (Cognitive Exercise Therapy Approach Questionnaire - BETY-BQ) Quality of life (Short Form-12) Study findings are expected to provide evidence for the effectiveness of exergame applications as an enjoyable rehabilitation approach for individuals with fibromyalgia.

DETAILED DESCRIPTION:
Fibromyalgia (FM) is a chronic disorder characterized by widespread pain, tenderness in specific musculoskeletal regions, fatigue, sleep disturbances, headaches, cognitive dysfunction, muscle weakness, postural instability, altered gait, and an increased risk of falls. Exercise has been reported to be one of the most effective non-pharmacological treatments for FM, and various types of exercise have been proposed. However, the evidence regarding which type of exercise provides optimal benefit remains limited.

Recently, exergame-based exercises - video game-assisted physical activities that combine interactive gaming with exercise - have gained attention as a novel and motivating rehabilitation approach. These programs have been shown to enhance adherence and engagement in different populations, including healthy adults, older individuals, and patients with neurological and musculoskeletal conditions. Nevertheless, research on the use of exergames in individuals with fibromyalgia is scarce, and no studies have been identified that use the Nintendo Switch Ring Fit Adventure game in this population.

This randomized clinical trial aims to compare the effects of an exergame-based exercise program and a home-based exercise program in women diagnosed with fibromyalgia. Participants will be randomly assigned to one of two groups: (1) the exergame group, performing supervised exercises using Ring Fit Adventure twice a week for four weeks, and (2) the home-based exercise group, performing a physiotherapist-prescribed home exercise program twice a week for four weeks.

All participants will be evaluated at baseline and after the 4-week intervention period, and reassessed following a 4-week detraining phase. Data obtained from this study will contribute to understanding the effects of exergame applications on pain, balance, functional mobility, and psychosocial outcomes in women with fibromyalgia. The results are expected to provide evidence supporting the use of exergame-based exercises as an enjoyable and effective approach within rehabilitation programs for individuals with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 30 and 70 years, which is an age range in which fibromyalgia (FM) is more prevalent;
* Having a diagnosis of fibromyalgia;
* Being willing to participate in the study and signing the informed consent form;
* Meeting the 2016 American College of Rheumatology (ACR) diagnostic criteria, defined as a Widespread Pain Index (WPI) ≥ 7 and a Symptom Severity Scale (SSS) score ≥ 5, or WPI = 4-6 and SSS ≥ 9.

Exclusion Criteria:

* Pregnancy or breastfeeding
* Any known advanced pathology related to the locomotor system that contraindicates physical activity (such as arthritis, osteoarthritis, or uric acid disorders)
* Epilepsy
* History of severe headache
* Neurological disorder
* Peripheral neuropathy
* Known severe cardiovascular disease (such as endocranial hypertension, uncontrolled arterial hypertension, heart failure, or presence of a pacemaker)
* Orthopedic disorders of the upper or lower extremities that prevent participation in physical activity
* Rheumatologic disease other than fibromyalgia
* Pneumothorax
* Neoplasia
* Surgery within the last four months
* Severe psychiatric illness (such as uncontrolled depression and anxiety, personality disorders, dementia, or cognitive impairments related to substance abuse)
* Diagnosis of alcohol dependence or use of psychoactive drugs or narcotics
* Participation in any physical activity program within two months prior to the start of the study
* Body mass index (BMI) greater than 29.9

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-05 (Estimated)

PRIMARY OUTCOMES:
Revised Fibromyalgia Impact Questionnaire | Assessed at baseline, post-intervention (4 weeks), and at 8-week follow-up
  The Revised Fibromyalgia Impact Questionnaire will be used to assess the impact of fibromyalgia (FM) on patients. The questionnaire consists of 21 items. All items are based on an 11-point numerical rating scale ranging from 0 to 10, where 10 indicates the worst possible condition. It comprises three domains: function, overall impact, and symptoms. The total score for the function domain (range 0-90) is divided by 3; the overall impact domain (range 0-20) is left unchanged; and the total score for the symptom domain (range 0-100) is divided by 2. The overall Revised Fibromyalgia Impact Questionnaire score is the sum of these three domain scores.
Fibromyalgia Severity Scale | Assessed at baseline, post-intervention (4 weeks), and at 8-week follow-up
  The Fibromyalgia Severity Scale is calculated by summing the scores of the Widespread Pain Index (WPI) and the Symptom Severity Scale (SSS). The maximum total score is 31 (19 + 12 = 31). A total score below 12 is generally not considered indicative of fibromyalgia.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | Assessed at baseline, post-intervention (4 weeks), and at 8-week follow-up
  The Visual Analog Scale is a 100-mm horizontal line used to assess pain intensity. Participants are asked to mark a point on the line that represents their current level of pain. A score of 0 indicates "no pain," while 100 represents "the worst pain imaginable." The measurement is recorded in centimeters.
30-Second Sit-to-Stand Test | Assessed at baseline, post-intervention (4 weeks), and at 8-week follow-up
  A 45 cm-high armless chair and a stopwatch will be used. Participants sit upright with feet flat on the floor and arms crossed over the chest. On the "start" command, they stand up and sit down as many times as possible within 30 seconds. The total number of full stands is recorded as the score. The chair will be stabilized against a wall, and each participant will receive verbal instructions, a demonstration, and 2-3 practice trials.
Timed Up and Go Test | Assessed at baseline, post-intervention (4 weeks), and at 8-week follow-up
  Functional mobility will be assessed by measuring the time taken to stand up from a chair, walk 3 meters, turn around, and sit down again. Three trials will be performed, and the best time recorded.
Single-Leg Stance Test | Assessed at baseline, post-intervention (4 weeks), and at 8-week follow-up
  Static balance will be evaluated by asking participants to stand on one leg with arms crossed at the chest, eyes open, and without support. The duration of maintaining the position will be recorded in seconds. The test will stop at 120 seconds and will be performed bilaterally (Akıl et al., 2020; Springer et al., 2007).
Berg Balance Scale | Assessed at baseline, post-intervention (4 weeks), and at 8-week follow-up
  The scale consists of 14 tasks scored from 0 to 4, with a maximum total of 56 points. Scores of 0-20 indicate balance impairment, 21-40 acceptable balance, and 41-56 good balance.
Cognitive Exercise Therapy Approach Scale (BETY-BQ) | Assessed at baseline, post-intervention (4 weeks), and at 8-week follow-up
  This 30-item questionnaire, scored on a 5-point Likert scale (0-4), assesses biopsychosocial impact. Higher scores indicate greater impact.
Short Form-12 (SF-12) | Assessed at baseline, post-intervention (4 weeks), and at 8-week follow-up
  The SF-12, a short version of the SF-36, assesses physical and mental health over the past four months. Higher scores reflect better health status. The Turkish version has been validated.

CONTACTS AND LOCATIONS:
Overall Officials: Gülhan Fetin, PT, Principal Investigator — Halic University
Locations (1):
- Halic University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No